CLINICAL TRIAL: NCT06219135
Title: Evaluation of the Performance of the IDBIORIV Method in Pathogen Identification and Antibiotic Susceptibility Testing in Patients With Sepsis
Acronym: IDBIORIV
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0542; 2023-A01260-45 (Other: ANSM)
Record Dates: First submitted 2023-12-06; First posted 2024-01-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Sepsis; bacteria; microbiology diagnosis method; identification; resistance; antibiotic susceptibility testing; virulence
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For each participant, a strain of the detected pathogen will be stored at the Institut des Agents Infectieux of the Centre de Biologie and Pathologie Nord of the Hôpital de la Croix Rousse 69004 Lyon.
  In option, for adult patients with Bacteraemia (bacteraemia group only), a blood sample will be drawn at visit H24-48 and J30. Analysis will be done at Laboratoire Commun de Recherche Hospices Civils de Lyon-bioMérieux, 69310 Pierre Bénite
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Contamination: Patients with a positive blood culture due to contamination microorganism
  Interventions: Other: no intervention - Contamination group
- Bacteraemia: This group includes all adults and children with a positive blood culture due to pathogen microorganism
  Interventions: Biological: blood sample - Bacteraemia group
- Emergency: Emergency Room Patient's with a positive blood culture due to pathogen and/or contamination microorganism
  Interventions: Other: no intervention - Emergency group

INTERVENTIONS:
Other: no intervention - Contamination group — there is no intervention for this group of patients
  Groups: Contamination
Biological: blood sample - Bacteraemia group — for adult patients, in optional, blood sample will be taken. 27,5 ml of blood at H24-48 after inclusion and 5 ml of blood at day 30
  Groups: Bacteraemia
Other: no intervention - Emergency group — there is no intervention for this group of patients
  Groups: Emergency

SUMMARY:
Sepsis is a disruption of homeostasis in the human body in response to bloodstream infection and is associated with a high risk of mortality.

Worldwide, sepsis is affecting approximately 30 million people and resulting in six million deaths.

Blood culture is a specific blood sample used to identifying microbial agent (bacterium or yeast) and determine the sensitivity of these microorganisms to antibiotics and antifungals.

Any delay in identifying the microorganism and/or determining the AST (antibiotic susceptibility testing) has a direct impact on the administration of appropriate antibiotic treatment and, consequently, on mortality of the patient. The faster the diagnosis, the faster the antibiotic treatment will be adapted, the higher the survival rate/probability of patients, and the lower the ecological impact.

In routine, clinical microbiology laboratories currently use 2 automatized techniques: MALDI-TOF MS® for microorganisms identification and VITEK2® method for AST determination.

Based on a proteomic approach, the IDBIORIV method is a rapid method (90 minutes) in comparison of current methods (24/48 hours) able to identifying a large panel of 113 pathogens and determine the antibiotic resistance profile of 49 species for 4 classes of antibiotics (Beta-lactams, Aminosides, Glycopeptides, Colistin).

The main objective of this study is to evaluate the performance of the IDBIORIV method in pathogen identification and antibiotic susceptibility testing in comparison with current methods of analysis of positive blood cultures used at the microbiology laboratory of the Hospices Civils de Lyon, in a real clinical situation, over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child patient
* Hospitalized in one of the departments registered with Hospices Civils de Lyon
* Showing signs of infection
* Confirmed by a 1st positive blood culture
* Patient or close relative (trustworthy person or family member) or holder of parental authority who has given his or her non-objection after receiving the information note

Exclusion Criteria:

* Patients under court protection
* Patients under guardianship or curatorship

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will focus on adult and pediatric patients hospitalized in 23 clinical departments of the Hospices Civils de Lyon and presenting a first positive blood culture detected on the microbiology laboratory of the Institut des Agents Infectieux.
Sampling Method: Non-Probability Sample
Enrollment: 1372 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The IDBIORIV method will be compared with the current routine methods present in the Hospices Civils de Lyon. The sensitivity and specificity of the IDBIORIV method will be evaluated using the Identification (ID) results of a positive blood culture for a | 24 Hours to 48 Hours after inclusion
  Reference technique used = Vitek MS ® (MALDI-ToF) bioMérieux.
The IDBIORIV method will be compared with the current routine methods present in the Hospices Civils de Lyon. The sensitivity and specificity of the IDBIORIV method will be evaluated using AST results. Reference technique = Vitek 2® bioMérieux | 24 Hours to 48 Hours after inclusion
  The performance of the IDBIORIV method for in vitro diagnosis of antibiotic-resistant/susceptible status will be evaluated for each "species-antibiotic" pair and "species-antibiotic group" of interest.
  Sensitivity will be calculated as the proportion of pairs diagnosed as resistant using the IDBIORIV method among pairs diagnosed as resistant using AST.
  Specificity will be calculated as the proportion of pairs diagnosed as sensitive with the IDBIORIV method among pairs diagnosed as sensitive with AST.

CONTACTS AND LOCATIONS:
Overall Officials: François VANDENESCH, Pr, Study Director — Hospices Civils LYON
Locations (8):
- France (8):
  - Femme Mère enfant Hospital, Bron
  - Femme Mère Enfant Hospital, Bron
  - Louis Pradel Hospital, Bron
  - Pierre Wertheimer Hospital, Bron
  - Edouard Herriot Hospital, Lyon
  - Croix Rousse Hospital, Lyon
  - Lyon Sud Hospital, Pierre-Bénite
  - Charpennes Hospital, Villeurbanne